CLINICAL TRIAL: NCT02403960
Title: The Effect of a Streptococcus Probiotic in Periodontal Therapy: a Randomized Controlled Trial
Brief Title: Probiotic Use in Chronic Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Onur Ozcelik, Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CukurovaU3
Record Dates: First submitted 2015-03-16; First posted 2015-03-31 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic (Active Comparator): The participants of the probiotic group were asked to let a probiotic tablet dissolve on their tongue 2 times a day for 3 months.
  Interventions: Dietary Supplement: probiotic
- placebo (Placebo Comparator): The participants of the control group were asked to let a placebo tablet dissolve on their tongue 2 times a day for 3 months.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: probiotic — the patients used probiotic tablets in addition to scaling and root planning
  Arms: probiotic
Dietary Supplement: placebo — the patients used placebo tablets in addition to scaling and root planning
  Arms: placebo

SUMMARY:
Aim: to evaluate the additional effects of the 12 weeks usage of a Streptococcus containing probiotic tablet after scaling and rootplaning compared to a placebo tablet.

Materials and methods: 48 periodontitis patients were included in this double-blind, placebo-controlled trial. After scaling and rootplaning, they were given patients used either a placebo (SRP) or probiotic tablet (SRP + P), 2 times a day for 12 weeks. Clinical and microbiological parameters were studied recorded up to 24 weeks after scaling and rootplaning.

DETAILED DESCRIPTION:
Materials and methods This double-blind, placebo-controlled, randomized (1:1 ratio) controlled trial with two parallel arms involved 48 patients with advanced adult periodontitis. They were recruited at the periodontology department of the Cukurova university, Turkey. All patients referred for periodontal treatment were screened for eligibility.The project was approved by the ethical committee for clinical trials of the Cukurova University in Turkey with number . No changes in the trial design were made after approval by the Ethical Committee.

Sample size calculation and randomization Power analysis prior to the start of the study was difficult since no previous randomized controlled trials on this study product were available. The sample size was determined. Pocket probing depth was taken into account, with an expected difference of 0.82mm and a standard deviation of 0.61mm. It was calculated that 10 patients were needed in each group to provide 80% power with an alpha of 0.05 . Despite this low number and taking into consideration studies comparing the adjunctive effect of antibiotics to scaling and rootplaning, it was decided to include 24 patients in each group.

Randomization of the patients was done by block randomization . The study coordinator distributed the coded bottles to the examiner at baseline, 4 weeks and 8 weeks visit. Except for the study coordinator, all patients and study personnel were blinded to the study group allocation. Before sending the data to the biostatistician, the code was broken to group the patients to the proper groups.

Treatment protocol Patients fulfilling the eligibility criteria were asked to participate in the study and after approval to sign an informed consent. Baseline examination included full-mouth probing pocket depth , gingival recession and bleeding on probing measured at six sites per tooth. Additionally the plaque en gingival indexes were noted. The full-mouth plaque index was recorded.After baseline periodontal examination and microbial analysis, an oral hygiene instruction was given (toothbrush, interdental brush). Initial periodontal therapy consisted of a full-mouth one-stage disinfection approach . All clinical procedures were performed by the same periodontist . The patient was asked to rinse for 2 minutes with a 0.12% chlorhexidine solution without alcohol . Scaling and rootplaning were performed on 2 consecutive days using an ultrasonic scaler under 0.12% chlorhexidine irrigation and with hand instruments. All mucosal surfaces were afterwards disinfected and the tongue was brushed for 1 minute. Besides, the participants were randomized over the 2 treatment groups: control or probiotic group.The participants of the probiotic group were asked to let a probiotic tablet dissolve on their tongue 2 times a day for 3 months. The participants in the control group were asked to do the same with a placebo tablet. All patients were instructed to use the tablets after brushing their teeth in the morning and in the evening. The probiotic and placebo tablets were identical in shape, texture, taste and composition except that Streptococcus were added for the probiotic tablet. All patients were supplied with the same toothpaste . It was asked not to use any probiotic containing products during the course of the study. Neither was it allowed to use drugs with anti-inflammatory properties, chlorhexidine or other mouthrinses during the study.

At designated time points, follow-up visits were planned. 30 days and 60 days after initiation of the therapy clinical evaluation and microbial analysis were performed. 90 days and 180 days after the initial treatment all baseline parameters were recorded .

Outcomes variables of interest Primary outcome measures The primary response variable was Probing pocket depth. All examinations were performed with a North Carolina periodontal probe .

Secondary outcome measures The secondary response variables were recession, clinical attachment level , Bleeding, Gingival index, Plaque index and microbial parameters.

Sub-analyses were performed on these outcome variables taking into account the initial Pocket. A pocket was considered moderate if its initial Pocket was between 4 and 6 mm and deep if ≥7 mm. "Risk for disease progression" was defined at patient level. The "need for surgery" outcome measure was calculated. A site was considered as "in need for surgery" if the Pocket was ≥6 mm or 5 mm and Bleeding positive. A tooth was considered in need for surgery if it had at least one site in need for surgery. A patient was considered in need or surgery if at least one tooth was in need for surgery.

Microbiological samples were collected of supragingival and subgingival plaque, saliva and the tongue. Pooled supragingival plaque samples were taken with the aid of curettes at the four single-rooted teeth with the deepest initial pocket in each quadrant. Before sampling, the sites were isolated from saliva with the aid of cotton rolls and then dried with compressed air. All supragingival plaque from these sites was dispersed. Samples were dispersed using a vortex mixer and immediately frozen at -20°C until analysis. On the same teeth pooled subgingival plaque samples were collected per site. After 10 s, the samples were transferred to a sterile Eppendorf tube, as described Saliva samples were obtained by collecting unstimulated saliva in a sterile cup. Finally the biofilm of the tongue was collected with a cotton swab. These were wiped 10 times over the tongue starting from the tongue dorsum.

Processing of the microbial samples After finishing the study, the frozen samples were send on dry ice to the department of Periodontology , these were immediately frozen at -80°C upon arrival. each sample was later defrosted and centrifuged at 13.000g. Bacterial DNA was extracted . A quantitative assay was performed to quantify certain bacteria.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were:

1. healthy, non-institutionalized male or female patients,
2. at least 35 years of age,
3. a minimum of 3 natural teeth in every quadrant and
4. previously untreated moderate to severe periodontitis

Exclusion Criteria:

Exclusion criteria were:

1. received antibiotics for any purpose within 6 months prior to entering the study or suffering from a disease condition that would typically require antibiotic prophylaxis before dental treatment,
2. a history of diabetes, rheumatic fever, liver or kidney disease, neurological deficiencies, or use of medication which may affect periodontal tissue (for example: phenytoin, cyclosporin, chronic use of non-steroidal anti-inflammatory drugs),
3. pregnancy,
4. acute oral lesions or necrotizing ulcerative periodontitis and
5. dental personnel

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
probing pocket depth | 24 weeks

SECONDARY OUTCOMES:
Recession | 24 weeks
  Recession as measured in millimeters.
clinical attachment level | 24 weeks
  clinical attachment level as measured in millimeters
Bleeding on probing | 24 weeks
  Bleeding as measured in presence or absence of bleeding on probing the sulcus
Gingival Index | 24 weeks
Plaque Index | 24 weeks
microbial counts of bacteria | 24 weeks
  microbial counts as measured in colony forming units

CONTACTS AND LOCATIONS:
Overall Officials: Onur Ozcelik, Study Chair — CU
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

REFERENCES:
- [Derived] Laleman I, Yilmaz E, Ozcelik O, Haytac C, Pauwels M, Herrero ER, Slomka V, Quirynen M, Alkaya B, Teughels W. The effect of a streptococci containing probiotic in periodontal therapy: a randomized controlled trial. J Clin Periodontol. 2015 Nov;42(11):1032-41. doi: 10.1111/jcpe.12464. Epub 2015 Nov 29. PMID 26427036